CLINICAL TRIAL: NCT00076271
Title: Evaluation and Treatment of Pediatric, Developmental and Genetic Eye Diseases
Brief Title: Evaluation and Treatment of Pediatric, Developmental, and Genetic Eye Diseases
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040039; 04-EI-0039
Record Dates: First submitted 2004-01-16; First posted 2004-01-19 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-10-28

CONDITIONS: Eye Diseases
Keywords: Strabismus; Cataract, Pediatric; Optic Nerve Anomaly; Coloboma; Evaluation and Treatment; Pediatric Ophthalmology; Genetic Eye Disease; Nystagmus; Pediatric Eye Disease; Developmental Eye Condition; Cataract; Juvenile Glaucoma; Eye Movement Disorder
MeSH Terms: conditions — Eye Diseases; Strabismus; Cataract; Coloboma; Nystagmus, Pathologic; Hydrophthalmos; Ocular Motility Disorders

SUMMARY:
This study will evaluate and treat children or adults with inherited or developmental eye conditions. It will allow specialists in pediatric ophthalmology, genetic ophthalmology, and ocular motility at the National Eye Institute (NEI) to learn more about the course of various pediatric, genetic, developmental, and eye movement diseases thorough long-term observation and treatment. It will also serve as the first step in determining the eligibility of patients who may wish to enroll in other NEI clinical research studies or undergo standard eye treatments.

Children with eye conditions, especially inherited or developmental conditions, and adults with eye disorders that began in childhood or that likely have a genetic or developmental component may be eligible for this study. Participants will undergo some or all of the following procedures:

* Medical history, including family history.
* Physical examination and possibly routine blood tests, x-rays tests, standard eye movement recordings, questionnaires, and specialized procedures when needed.
* Complete eye examination, including vision test, visual perception, eye pressure (if possible), dilation of the pupils to examine the back of the eye (lens, vitreous, and retina).
* Photographs of the eyes.
* Oculography (eye movement recordings) in patients for whom testing will aid in diagnosis. This test is done either with goggles placed over the eyes or with a contact lens placed on each eye. When the goggles or lenses are in place, the subject looks at a series of red targets on a computer screen.
* Electroretinography (ERG) in patients with suspected retinal degeneration. This is a test of the electrical function of the eyes. Before the test, patients sit in a dark room for 30 minutes with their eyes patched. A small electrode (silver disk) is taped to their forehead. The eye patches are then removed, the eyes are numbed with drops, and contact lenses are placed in the eyes. The contact lenses sense small electrical signals generated by the retina when lights flash. During the ERG recording, the patient looks inside a large empty bowl. A light flashes, first in the dark and then with a light turned on inside the bowl. The test takes 1 hour or less.

Participants are followed up to 6 times a year for 3 years, depending on the diagnosis and treatment.

DETAILED DESCRIPTION:
The purpose of this protocol is to allow the pediatric ophthalmology, genetic ophthalmology, and ocular motility specialists at the National Eye Institute to gain additional knowledge of the course of various pediatric, genetic, developmental and ocular motility diseases. Heretofore, this spectrum of diseases will be referred to as pediatric ophthalmology diseases. We wish to evaluate the effects of standard treatments for these diseases, use non- or minimally-invasive technologies to understand the pathogenesis of these diseases, and to collect blood or other easily obtained biologic sample (e.g., urine, saliva, hair, cheek swab, or stool) for future laboratory studies on these diseases. The information gained from this protocol will also allow for the maintenance of populations of patients with specific pediatric eye diseases and strabismus that may be eligible for future protocols. In addition, by allowing for the care of patients with a spectrum of these diseases, the protocol will be valuable for the training of pediatric eye disease, ocular genetics, and ocular motility fellows. The pediatric, genetic, and eye movement specialists at the National Eye Institute will choose ophthalmology diseases based on the training and research needs of the NEI program. While the primary focus of this protocol is to study eye disease in children, adults who have a disease that began in childhood or who may have an inherited eye disease or are unaffected first-degree relatives may also be evaluated under this protocol.

This protocol is not designed to test any new treatments. Any evaluation of treatments under this protocol will be based on the standard-of-care for each patient's disease. All alternatives for evaluation and care will be reviewed with each patient and the patient's family.

Patients in this evaluation and treatment protocol will be evaluated for potential eligibility in any new NEI clinical trials or epidemiological protocols as they are developed. If eligible, patients may be asked to participate in a new protocol. However, they will not be required to enter any new protocol and their decision to participate will be entirely voluntary.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects will be able to enroll if they:

1. Are a pediatric patient, of any age, with ophthalmic conditions, especially inherited or developmental conditions, OR
2. Are an adult patient with an eye disorder that began in childhood or that is likely to have a genetic/developmental component, OR
3. Are an unaffected first-degree relative that we believe that will aid in our diagnosis or future research objectives, AND
4. Have the ability to understand and sign an informed consent OR have a legal parent/guardian with the ability to do the same.

EXCLUSION CRITERIA:

Subjects will not be eligible if they:

1. Are unable to follow-up as clinically indicated.
2. Have a severe systemic disease that compromises our ability to provide adequate examination and/or treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350
Dates: Start 2004-01-14; Study Completion 2008-10-28

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rocky Mountain Lions Eye Institute, Denver, Colorado
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Tang J, Gokhale PA, Brooks SE, Blain D, Brooks BP. Increased corneal thickness in patients with ocular coloboma. J AAPOS. 2006 Apr;10(2):175-7. doi: 10.1016/j.jaapos.2005.12.003. No abstract available. PMID 16678756
- [Background] Chang L, Blain D, Bertuzzi S, Brooks BP. Uveal coloboma: clinical and basic science update. Curr Opin Ophthalmol. 2006 Oct;17(5):447-70. doi: 10.1097/01.icu.0000243020.82380.f6. PMID 16932062
- [Background] Brooks BP, Meck JM, Haddad BR, Bendavid C, Blain D, Toretsky JA. Factor VII deficiency and developmental abnormalities in a patient with partial monosomy of 13q and trisomy of 16p: case report and review of the literature. BMC Med Genet. 2006 Jan 13;7:2. doi: 10.1186/1471-2350-7-2. PMID 16412230